CLINICAL TRIAL: NCT06996015
Title: Effects of SNAGs and Cognitive Behavior Therapy on Pain, Craniovertebral Angle and Disability in Patients With Non-Specific Neck Pain
Brief Title: Effects of SNAGs & CBT on Pain, Craniovertebral Angle & Disability in Non Specific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0154
Record Dates: First submitted 2025-03-10; First posted 2025-05-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain; Cognitive Behavior Therapy; Cervicalgia; Posture; Posterior Neck Pain; Neck Pain and Forward Head Posture
Keywords: snags; Non-Specific Neck Pain; Craniovertebral Angle; disability
MeSH Terms: conditions — Neck Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): Cognitive Behavioral Therapy will be delivered in 20-minute sessions using visual aids like videos, images, and pamphlets to explain cervical spine structure, biomechanics, pain pathways, and ergonomic practices. Techniques for managing flare-ups and maintaining good posture will be taught, ensuring active engagement and focus. A manual summarizing key points will be provided, and students will be encouraged to ask questions. Sessions will occur twice weekly for four weeks.
  Interventions: Other: Cognitive behavior therapy
- Cervical Stabilization Exercises (Active Comparator): Cervical Stabilization Exercises (CSE) will include bracing techniques in neurodevelopmental stages (supine, prone, quadrupedal, bipedal) with 10-second holds for 10 repetitions. Extremity ROM exercises will be done while maintaining spinal stability, progressing from 8 to 12 reps. Cervical isometric exercises will target multiple directions using elastic bands, with 10 reps and 6-10 second holds. Functional training with elastic resistance and exercise balls on unstable surfaces will also be incorporated, with 10 reps and 10-15 second holds. Sessions will occur twice weekly for four weeks.
  Interventions: Other: Cervical Stabilization Exercises

INTERVENTIONS:
Other: Cognitive behavior therapy — The treatment session will begin with a 10-minute conventional therapy, including a 5-minute hot pack applied to the cervical region and a 5-minute Myofascial Release (MFR) using skin rolling and cross-hand techniques to relax and stretch the fascia layers. This will be followed by a 10-minute application of Sustained Natural Apophyseal Glides (SNAGs), where the physiotherapist will guide the patient's active neck movements with accessory glides to improve joint ROM and reduce pain. Lastly, a 20-minute Cognitive Behavioral Therapy (CBT) session will include visual aids, explanations of cervical spine biomechanics, pain pathways, ergonomics, and posture management. Patients will receive manuals summarizing key points and be encouraged to engage actively. The 40-minute session will be conducted twice weekly for four weeks
  Arms: Cognitive Behavior Therapy
Other: Cervical Stabilization Exercises — The treatment session will last 40 minutes, twice a week for 4 weeks. It begins with a 10-minute conventional treatment: a 5-minute hot pack application to the cervical region followed by a 5-minute Myofascial Release (MFR) using the skin rolling technique. Natural wax will be applied for smooth strokes. MFR will engage all fascia layers with superficial strokes, progressing to deeper fascia using cross-hand stretch, depending on the pain tolerance.
  Next, SNAGs (Sustained Natural Apophyseal Glides) will be applied for 10 minutes. The patient, seated, will actively move the painful joint through its range of motion while the therapist applies a glide force. This will be repeated 10 times for 3 sets.
  Then session includes 20 minutes of Cervical Stabilization Exercises (CSE) with bracing in neurodevelopment stages (supine, prone, quadrupedal, bipedal), holding each position for 10 seconds. Isometric exercises and functional training with elastic bands and exercise balls follow.
  Arms: Cervical Stabilization Exercises

SUMMARY:
Non-specific neck pain is a prevalent condition causing discomfort, reduced craniovertebral angle, and disability. This randomized controlled trial will evaluate the combined effects of Sustained Natural Apophyseal Glides (SNAGs) and Cognitive Behavioral Therapy (CBT) on pain, posture, and function. Group A will receive SNAGs and CBT, while Group B will undergo SNAGs with cervical stabilization exercises, twice weekly for four weeks. Outcomes will include pain, craniovertebral angle, and disability, analyzed using SPSS.

DETAILED DESCRIPTION:
Non-specific neck pain is a common musculoskeletal disorder that will affect a significant portion of the population, leading to discomfort, reduced craniovertebral angle, and functional disability. While traditional physical therapy methods provide symptomatic relief, there is growing interest in integrating psychological interventions to address underlying factors contributing to chronic pain. This study will investigate the combined effects of Sustained Natural Apophyseal Glides (SNAGs) and Cognitive Behavioral Therapy (CBT) on pain reduction, craniovertebral angle improvement, and disability in patients with non-specific neck pain.

This study will be a randomized controlled trial involving -- patients diagnosed with non-specific neck pain. Participants will be randomly assigned into two groups. Both groups will receive conservative treatment, including a 5-minute hot pack application and 5 minutes of myofascial release. Subsequently, SNAGs will be administered for 10 minutes to both groups. Group A will receive an additional 20-minute session of Cognitive Behavioral Therapy (CBT) focusing on pain management strategies. In contrast, Group B will receive cervical stabilization exercises for 20 minutes. The intervention will be administered twice a week for four weeks. Pain intensity, craniovertebral angle, and disability will be measured at baseline and post-intervention using standardized assessment tools. Data analysis will be performed using SPSS version 25, with within-group and between-group comparisons to evaluate the efficacy of the interventions.

Existing studies focus on manual therapies and short-term outcomes but lack insights into the combined and sustained effects of SNAGs and CBT. This research aims to bridge that gap, exploring the physical and psychological dimensions of treatment to improve long-term function and patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-28 Years(20)
* Gender Group: Both male and female participants(20)
* Individuals with a Craniovertebral angle <53(20)
* Individuals having grade 2 neck pain according to KNGF Guidelines.(21)
* Individuals having localized pain or stiffness in spine or both combined between C3 and C7 without upper-limb radiculopathy(22)
* Individual who had not received any treatment for neck pain for the last 3 months will be included in the study.
* Patients willing to sign written consent form.

Exclusion Criteria:

* Those who had undergone spinal surgery(23)
* Neck pain caused by various pathologies (rheumatoid arthritis, ankylosing spondylitis, fracture, tumor, etc.)(23)
* Nerve root compression, (23)
* A positive vertebrobasilar artery test, (23)
* Severe radiculopathy,(23)
* Osteoporosis, or osteopenia(23)
* Long-term use of corticosteroids or anticoagulants (23)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
NPRS | 4th week
  Numerical Pain Rating Scale (NPRS) To determine the degree of pain that the patient will report, the Numeric Pain Rating Scale (NPRS) will be utilized. This scale consists of 11 points ranging from 0-10, where zero indicates no pain, five represents moderate pain intensity, and ten signifies severe pain intensity.
  An intraclass correlation value (ICC) of 0.67 indicated a moderate level of reliability for the NPRS (Numeric Pain Rating Scale), indicating a moderate level of consistency and stability in the scores obtained from the measurement tool.(24) NPRS have shown high test-retest reliability (r = 0.96 and 0.95, respectively) (19).
  The measurements for pain intensity will be recorded through this scale at baseline, and after 4 weeks of treatment
Neck Disability Index | 4th week
  To assess neck-related disability, a questionnaire called the Neck Disability Index (NDI) will be used. It consists of eleven things that address pain and regular tasks such personal care, lifting, reading, headaches, focusing, work status, driving, sleeping, and recreation.
  The intraclass correlation coefficient (ICC) for the NDI (Neck Disability Index) is 0.88, indicating very high reliability, indicating a high level of consistency and stability of scores obtained from the measurement tool.(24) It has been demonstrated that the NDI-U questionnaire can accurately assess neck impairment in Urdu-speaking individuals with chronic musculoskeletal neck pain (CMNP). Its two-factor structure and use of simple language make it easy for patients to understand, making it a suitable assessment tool in both clinical and research settings for patients population.(25)

SECONDARY OUTCOMES:
Craniovertebral Angle | 4th week
  Photogrammetric method (for Measuring Craniovertebral Angle):
  Neck pain is frequently brought on by the forward head posture, also referred to as the Craniovertebral Angle (CA). It is calculated using the angle created by a horizontal line going through the spinous process of C7 and a line originating from the tragus of the ear.
  According to intraclass correlation coefficient (ICC) values ranging from 0.88 to 0.98, photogrammetry in the sagittal plane is a trustworthy technique for determining forward head posture. This method has been utilized in several research studies to measure forward head posture.
  When used to evaluate cervical range of motion in the sagittal plane, the Kinovea software has also been demonstrated to have both intrarater and interrater reliability.
  This angle will be used to assess the degree of forward head posture in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Shaukat, TDPT, Principal Investigator — Riphah International University
Locations (1):
- Syeda Khatoon e Jannat Trust Hospital,, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No